CLINICAL TRIAL: NCT03442556
Title: PLATI-PARP: A Phase 2 Study of Induction Docetaxel and Carboplatin Followed by Maintenance Rucaparib in Treatment of Patients With Metastatic Castration Resistant Prostate Cancer With Homologous Recombination DNA Repair Deficiency
Brief Title: Docetaxel, Carboplatin, and Rucaparib Camsylate in Treating Patients With Metastatic Castration Resistant Prostate Cancer With Homologous Recombination DNA Repair Deficiency
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to insufficient funding
Sponsor: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9841; NCI-2018-00016 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9841 (Other: Fred Hutch/University of Washington Cancer Consortium); RG1717043 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2018-02-09; First posted 2018-02-22 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: ATM Gene Mutation; BRCA1 Gene Mutation; BRCA2 Gene Mutation; Castration Levels of Testosterone; Castration-Resistant Prostate Carcinoma; Homologous Recombination Deficiency; Prostate Carcinoma Metastatic in the Bone; PSA Level Greater Than or Equal to Two; PSA Progression; Stage IV Prostate Adenocarcinoma AJCC v7
MeSH Terms: interventions — Carboplatin; Docetaxel; rucaparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (docetaxel, carboplatin, rucaparib camsylate) (Experimental): INDUCTION: Patients receive docetaxel IV and carboplatin IV on day 1. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Patients receive rucaparib camsylate PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Docetaxel; Other: Laboratory Biomarker Analysis; Drug: Rucaparib Camsylate; Drug: Rucaparib

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP56976; Taxotere; Taxotere Injection Concentrate
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Rucaparib Camsylate — Given PO
  Other Names: 8-Fluoro-2-{4-[(methylamino)methyl]phenyl}-1,3,4,5-tetrahydro-6H-azepino[5,4,3-cd]indol-6-one ((1S,4R)-7,7dimethyl-2-oxobicyclo[2.2.1]hept-1-yl)methanesulfonic Acid Salt; C0-338; Rubraca; Rucaparib Phosphate
Drug: Rucaparib — Given PO
  Other Names: 283173-50-2; 6H-Pyrrolo(4,3,2-ef)(2)benzazepin-6-one; 8-Fluoro-1,3,4,5-tetrahydro-2-(4-((methylamino)methyl)phenyl)-

SUMMARY:
This phase II trial studies how well docetaxel with carboplatin followed by rucaparib camsylate works in treating patients with metastatic castration resistant prostate cancer (spread outside of prostate and resistant to testosterone suppression) with homologous recombination DNA repair deficiency. Chemotherapy drugs, such as docetaxel and carboplatin, work to stop the growth of cancer cells, by stopping them from dividing or spreading. Rucaparib camsylate may stop the growth of tumor cells with defects in the ability to repair mistakes in DNA by forcing additional errors so that the cancer cells cannot overcome the number of errors and will then die. Giving induction docetaxel and carboplatin followed by maintenance rucaparib camsylate may work better in treating patients with castration resistant prostate cancer.

DETAILED DESCRIPTION:
OUTLINE:

INDUCTION: Patients receive docetaxel intravenously (IV) and carboplatin IV on day 1. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients receive rucaparib camsylate orally (PO) twice daily (BID) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form (ICF) providing agreement to adhere to the dosing schedule, report for all trial visits and authorization, use and release of health and research trial information
* Histologically or cytologically confirmed adenocarcinoma of the prostate (excluding predominant small cell histology)
* Ongoing gonadal androgen deprivation therapy with gonadotropin-releasing hormone (GnRH) analogues, antagonists or orchiectomy; patients who have not had an orchiectomy must be maintained on effective GnRH analogue/antagonist therapy
* Castration resistant prostate cancer as defined by serum testosterone < 50 ng/ml and PSA level of at least 2 ng/ml that has risen on at least 2 successive occasions at least 1 week apart
* Presence of metastatic disease on bone or computed tomography (CT) scan

  * Evaluable disease progression by modified RECIST 1.1 (Response Evaluation Criteria in Solid Tumors)
  * Bone disease on bone scan
* Prior therapy with sipuleucel-T, abiraterone, enzalutamide, docetaxel, and/or cabazitaxel; there is no limit to the number of prior treatment regimens in the castration resistant setting, so long as prior therapy does not include platinum chemotherapy or a PARP inhibitor; prior platinum chemotherapy in the hormone sensitive setting is permitted, so long as it has been at least 6 months since last dose
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 1
* Life expectancy >= 12 weeks
* No prior malignancy is allowed except:

  * Adequately treated basal cell or squamous cell skin cancer or
  * In situ carcinoma of any site or
  * Other adequately treated malignancy for which the patient has been disease-free for at least one year (any prior chemotherapy is allowed)
* Documented evidence of at least ONE or MORE of the following:

  * Pathogenic mutation or inactivating alteration of a gene involved in homologous recombination repair in the tumor
  * Note, that if this alteration is identified in a circulating tumor deoxyribonucleic acid (ctDNA) assay, the variant-allele fraction must be > 20% to indicate relevance to predominant tumor clone

    * Mutation in one or more other genes involved in homologous DNA recombination repair in the tumor may be included at investigator's discretion
    * Homologous recombination repair deficiency by genomic signature in the tumor by BROCA-HR, Foundation One or equivalent assay
    * Presence of pathogenic or likely pathogenic germline mutation/variant in BRCA2, BRCA1, ATM or PALB2
  * Note: Germline mutations in other HR genes will be considered at investigator's discretion)
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (within 14 days of first dose of study drug)
* Platelets > 100 x 10^9/L (within 14 days of first dose of study drug)
* Hemoglobin >= 9 g/dL (within 14 days of first dose of study drug)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3 x ULN; if liver metastases, then =< 5 x ULN (within 14 days of first dose of study drug)
* Bilirubin =< 1.5 x ULN (< 2 x ULN if hyperbilirubinemia is due to Gilbert's syndrome) (within 14 days of first dose of study drug)
* Serum creatinine =< 1.5 x ULN or estimated glomerular filtration rate (GFR) >= 45 mL/min using the Cockcroft Gault formula (within 14 days of first dose of study drug)

Exclusion Criteria:

* Currently receiving active therapy for other neoplastic disorders
* Symptomatic and/or untreated central nervous system (CNS) metastases; patients with asymptomatic previously treated CNS metastases are eligible provided they have been clinically stable for at least 4 weeks
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness, active or symptomatic viral hepatitis or chronic liver disease
* Clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, or New York Heart Association (NYHA) class II-IV heart disease or cardiac ejection fraction measurement of < 35 % at baseline
* Treatment with an investigational therapeutic drug within 30 days of cycle 1
* Prior therapy with a PARP inhibitor (e.g., olaparib, talazoparib, veliparib, niraparib, rucaparib)
* Prior therapy with a platinum chemotherapy (e.g. cisplatin, carboplatin, oxaliplatin) in the castration resistant setting; (prior platinum chemotherapy in the hormone sensitive setting is permitted, so long as time since last dose is 6 months or greater)
* Active, ongoing toxicity (Common Terminology Criteria for Adverse Events [CTCAE] grade 2 or higher) from prior therapy
* Presence of dementia, psychiatric illness, and/or social situations limiting compliance with study requirements or understanding and/or giving of informed consent
* Pre-existing duodenal stent and/ or any gastrointestinal disorder or defect that would, in the opinion of the Investigator, interfere with absorption of rucaparib
* Any condition(s), medical or otherwise, which, in the opinion of the investigators, would jeopardize either the patient or the integrity of the data obtained

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-08-24 (Actual); Primary Completion 2025-06-04 (Actual); Study Completion 2025-06-04 (Actual)

PRIMARY OUTCOMES:
Radiographic progression free survival assessed by assessment using the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1/Prostate Cancer Working Group 3 (PCWG3) criteria | From first dose of docetaxel/carboplatin to the date of first objective evidence of radiographic progression (soft tissue or bone lesion) or death due to any cause, whichever occurs first, assessed up to 6 years

SECONDARY OUTCOMES:
Overall response rate (ORR) of measurable disease (PCWG3) (complete response or partial response) assessed by modified RECIST version 1.1 criteria | Up to 6 years
Prostate-specific antigen (PSA) nadir after induction | Up to 6 years
  Rate of confirmed PSA decrease from baseline, assessed by a local laboratory (PSA50 and PSA90)
PSA nadir after maintenance | Up to 6 years
  Rate of confirmed PSA decrease from baseline, assessed by a local laboratory (PSA50 and PSA90)
PSA response duration | From the date that a response (PSA decrease >= 50%) is first reported to the time that PSA progression is first documented, assessed up to 6 years
Time to PSA progression (PCWG3) | From first dose of docetaxel/carboplatin to the date that a >= 25% increase and absolute increase of >= 2 ng/mL above the nadir (or baseline value for patients who did not have a decline in PSA) in PSA was measured, assessed up to 6 years
  The increase must be confirmed by a second consecutive assessment conducted at least 3 weeks later.

CONTACTS AND LOCATIONS:
Overall Officials: Heather H. Cheng, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No